CLINICAL TRIAL: NCT04769778
Title: Renin Angiotensin System Blockade in Renal Transplant Patients With Presence of PECs in Urine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josep M Cruzado (Other)
Responsible Party: Sponsor-Investigator, Josep M Cruzado, Head of Nephrology, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRONE
Record Dates: First submitted 2021-01-07; First posted 2021-02-25 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Allograft Nephropathy
Keywords: renin angiotensin; kidney transplant; PEC's
MeSH Terms: interventions — Valsartan; Tablets

STUDY DESIGN:
Intervention Model Description: Treatment with valsartan versus no treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valsartan (Experimental): Treatment with valsartan
  Interventions: Drug: Valsartan 80Mg Oral Tablet
- no treatment (No Intervention): no treatment received

INTERVENTIONS:
Drug: Valsartan 80Mg Oral Tablet — treatment with 80mg /day of valsartan
  Arms: Valsartan

SUMMARY:
By means of a personalized medicine strategy, investigators are going to evaluate if the treatment with an angiotensin II receptor antagonist (ARAII) in renal transplant patients with the presence of renal progenitor cells (PECs) in the urine is able to prevent the expected loss of glomerular filtration (GFR) observed in this subgroup of patients. In addition, investigators intend to deepen the mechanisms of glomerular damage and glomerular repair involved in the process of chronic allograft damage.

DETAILED DESCRIPTION:
A randomized, double-blind clinical trial will be performed in renal transplant patients in month 6 post-transplant, at the time of protocol renal biopsy. After verifying the inclusion and exclusion criteria, informed consent will be obtained. Patients with urinary PECs will be randomized to 80 mg of valsartan vs. placebo (sample size calculated for a superiority study, 45 patients per group). Patients without PECs in urine will be followed according to usual clinical practice. The follow-up will be up to 2 years post-transplant. At baseline (6 m post-transplant) and at 2 years the GFR will be measured by means of iohexol clearance (main variable) and, in addition, we will analyze safety variables such as patient and graft survival and RAGIs. By means of morphometry techniques on renal biopsy and by measuring the renal cortical volume by high resolution CT, the number of glomeruli will be determined, which in turn, will allow to calculate the SN-GFR. Finally, in 5 patients per study group and in 5 controls, PECs of renal tissue will be isolated by means of laser microdissection techniques to perform single-cell RNA sequencing techniques to assess the molecular pathways involved in the glomerular damage and repair process and how the RAAS blockade modifies such molecular pathways.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Stable renal function understood as a variation of eGFR of less than 15% in the last 3 months
* Immunosuppression maintenance based on tacrolimus and MMF / MPA

Exclusion Criteria:

* Chronic active infection by HCV, HBV, HIV.
* Treatment with inhibitors of the renin angiotensin system.
* Double kidney transplant or combined with another organ.
* Immunosuppression of maintenance other than tacrolimus and MMF / MPA.
* eGFR <20 ml / min / 1.73m2.
* History of allergy or intolerance to inhibitors of the renin angiotensin system.
* Physically fertile women who plan to become pregnant, are pregnant and

  / or breast-feeding, or who do not want to use effective contraception during their participation in the study.
* Any other medical condition that, in the opinion of the investigator, based on the counting or review of clinical records, could affect the completion of the study, including, but not limited to, visual problems or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
prevention of fall of glomerular filtration rate | 12 months
  To assess whether treatment with an angiotensin II receptor antagonist (AIIRA) prevents the fall of glomerular filtration in the subgroup of kidney transplant patients with presence of PECs in urine.

SECONDARY OUTCOMES:
SN-GFR | 12 months
  Compare the SN-GFR (nephron glomerular filtration rate)
Single cell RNA sequencing | 12 months
  Carry out single cell RNA sequencing studies using cell microdissection techniques of PEC cells isolated from renal biopsies performed at 6 and 24 m after transplantation in patients without uPECs and in patients with uPECs included in the therapeutic intervention study. These studies will allow us to know the changes of gene expression in PECS cells that can be associated with the favorable response in treated or untreated patients.
podocyturia | 12 months
  To determine the influence of the treatment on podocyturia and the preservation of the number of podocytes at 2 years post transplant.
graft survival | 12 months
  Evaluate the influence of treatment on graft survival
patient survival | 12 months
  Evaluate the influence of treatment on patient survival and proteinuria.
Chronic Glomerular Lessions | 12 months
  Evaluate the influence of treatment on number of participants with chronic glomerular lesions.
Suspected Unexpected Serious Adverse Reaction (SUSAR) reporting unexpected serious adverse reactions) | 12 months
  Evaluate the safety of the treatment on the number of patients with Suspected Unexpected Serious Adverse Reaction (SUSAR) reporting unexpected serious adverse reactions) unexpected adverse reactions) and rate of treatment discontinuations.
Proteinuria | 12 months
  Evaluate the influence of treatment on measure of proteinuria

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Department. Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain